CLINICAL TRIAL: NCT06638034
Title: Diagnosis of Metastatic Tumors on 68Ga-FAPI-RGD PET-CT and Radioligand Therapy
Brief Title: Diagnosis of Metastatic Tumors on 68Ga-FAPI-RGD PET-CT and Radioligand Therapy With 177Lu-FAPI-RGD
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Zhaohui Zhu, Clinical Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-FR-TRT
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: FAP- Expressing Positive Tumors; RGD- Expressing Positive Tumors
MeSH Terms: interventions — 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-FAPI-RGD PET/CT for scan and 177Lu-FAPI-RGD for therapy (Experimental): All patients diagnosed with metastatic tumors underwent 68Ga-FAPI-RGD PET/CT scan. If the PET/CT showed high FAPI expression in tumor lesions of some patients, they would intravenously injected with the dose about 2.22-3.33 GBq (60-100 mCi) of 177Lu-FAPI-RGD for therapy.
  Interventions: Drug: 68Ga-FAPI-RGD for PET / CT scan and 177Lu-FAPI-RGD for therapy

INTERVENTIONS:
Drug: 68Ga-FAPI-RGD for PET / CT scan and 177Lu-FAPI-RGD for therapy — Patients with positive results were screened with 68Ga-FAPI PET / CT, and 2.22-3.33GBq(60mci-100mCi) 177Lu-FAPI-RGD was injected intravenously for therapy after contraindications were excluded and informed consent was signed.

SUMMARY:
FAP and RGD are overexpressed in many tumor tissues. This study is intended to conduct preliminary clinical transformation and internal irradiation dosimetry research on 177Lu-FAPI-RGD--a new dual-targeted 177Lu therapeutic drug for the first time in the world.

DETAILED DESCRIPTION:
Fibroblast activation protein (FAP) and RGD are serine peptidase on the surface of tumor associated fibroblasts. It has special biological characteristics and stable genome. They are usually not expressed or expressed at a low level in the resting tissues of normal adults, but it is highly expressed in diseases related to tissue repair and matrix reconstruction,Receptor imaging with a single target also has some limitations in clinical application. For example, not all diseased cells express a large amount of single receptor on the surface, which greatly affects the judgment of the nature of the lesion. The dual-target molecular imaging based on FAP expressed in the lesion site and integrin αvβ3 receptor highly expressed on the surface of the lesion neovascularization will overcome the above limitations and make full use of the advantages of the dual-target molecular imaging, which will greatly assist the diagnosis of malignant tumors and used to 177Lu PRRT. We'll try to assess the safety and therapeutic response to 177Lu-FAPI-RGD in patients with metastatic tumors in human.

ELIGIBILITY:
Inclusion Criteria:

* confirmed treated or untreated metastatic tumors patients;
* 68Ga-FAPI PET/CT and 18F-FDG PET/CT within two weeks;
* signed written consent.

Exclusion Criteria:

* pregnancy;
* breastfeeding;
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
tandarStandardized uptake value of 177Lu-TATE-RGD in normal organs and tumors. | through study completion, an average of half-year
  The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake value at each time point in normal organs and tumors will be measured.
Adverse events collection | through study completion, an average of 2 months
  Adverse events within 2 months after the injection and scanning of patients will be followed and assessed.

SECONDARY OUTCOMES:
SUVmax, SUVmean, lesion-based analysis | through study completion, an average of 1 year
  Sensitivity and Specificity of 68Ga-FAPI PET/CT for metastatic tumors in comparison with 18F-FDG PET/CT, including some semi-quantative quota for lesion-based analysis, such as SUVmax, SUVmean

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Science & Peking Union Medical College Hospital, Beijing, Beijing Municipality, China